CLINICAL TRIAL: NCT06151275
Title: Factors Predict Difficult Colonoscopy Before the Procedure: Prospective Registry Study
Status: Completed | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Burak Dincer, Principal investigator, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: 30.05.2023-3951
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Colonoscopy
Keywords: Colonoscopy; Constipation; Cecal intubation time
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Colonoscopy: 18-95 years old patients apply our endoscopy unit for colonoscopy will be included in our study. Patients that have colonic resection history will be excluded from study.

SUMMARY:
In this study, the investigators aim to evaluate the relationship between cecal intubation time during colonoscopies and factors such as the patient's age, body mass index, history of constipation, Wexner constipation score, antidepressant use, and previous abdominal surgery. The objective is to assess factors that may predict longer cecal intubation times, especially in difficult colonoscopies. Prior to the procedure, informed consent will be obtained from patients scheduled for colonoscopy in the surgical endoscopy unit, and relevant information will be recorded. During the procedure, data will be collected, including cecal intubation time, if ileal intubation is performed, and the total procedure time.

DETAILED DESCRIPTION:
This study is designed as a prospective single-center registry study and has been approved by the Ethics Committee of Sisli Hamidiye Etfal Training and Research Hospital on May 30, 2023. The inclusion criteria for study involve patients scheduled for colonoscopy in surgical endoscopy unit who have not undergone colorectal surgery. Following informed consent obtained from patients before colonoscopy, data forms prepared by investigators will be completed, evaluating patients' age, height, weight, body mass index, colonoscopy indication, antidepressant use, and history of abdominal surgeries. Additionally, the Wexner constipation score will be calculated for each patient.

The time taken to reach the cecum and, if intubated, the ileum, from the initial insertion of the endoscope in colonoscopy, as well as the total procedure time, will be recorded using a chronometer. Patients with inadequate bowel preparation preventing cecal intubation will be excluded from the study. The collected data will be analysed to assess factors prolonging cecal intubation time and, if possible, to identify predictors for difficult colonoscopy before procedure.

ELIGIBILITY:
Inclusion Criteria:

* 18-95 years old, admitted for colonoscopy

Exclusion Criteria:

* Colonic resection history

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients that admit for colonoscopy to Sisli Hamidiye Etfal Research and Training Hospital
Sampling Method: Non-Probability Sample
Enrollment: 915 (Actual)
Dates: Start 2023-06-07 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
Cecal intubation rate | During the colonoscopy
  The rate of reaching the cecum in all colonoscopies performed
Ileal intubation rate | During the colonoscopy
  The rate of reaching the terminal ileum in all colonoscopies performed
Cecal intubation time | During the colonoscopy
  Time for reaching caecum starting from endoscope insertion, this time will recorded by chronometer and recorded as minutes
Ileal intubation time | During the colonoscopy
  Time for reaching ileum starting from endoscope insertion, this time will recorded by chronometer and recorded as minutes

SECONDARY OUTCOMES:
Adenoma detection rate | During the colonoscopy
  The rate at which endoscopists find one or more adenoma during colonoscopies

CONTACTS AND LOCATIONS:
Overall Officials: Burak Dincer, MD, Principal Investigator — Sisli Hamidiye Etfal Training and Research Hospital
Locations (1):
- Sisli Hamidiye Etfal Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No